CLINICAL TRIAL: NCT06782412
Title: Multicenter Validation Trial of [18F]AlF-FAPI-74 for PET Imaging of Cancer-associated Fibroblasts Through Fibroblast Activation Protein Inhibitors (FAPI) in Different Tumor Types
Acronym: FAPIDO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Principal Investigator, Christophe Deroose, Prof. Dr., Head of Clinic Nuclear Medicine, UZ Leuven - Full Professor, KU Leuven, KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S67792; 2024-512059-19 (EudraCT Number)
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Oesophageal Cancer; Gastric Cancer; Pancreatic Ductal Adenocarcinoma; FAP; Oncology; Oncologic Disorders
Keywords: Oesophagogastric adenocarcinoma; Pancreatic ductal adenocarcinoma; Clinically challenging situations; [18F]-FDG; [18F]-FAPI-74; [18F]AIF-FAPI-74; Positron emission tomography; PET; Nuclear imaging; Oncology; Prospective
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, multicenter, multi-cohort, interventional phase II/III trial.
  The three cohorts are: Oesophagogastric adenocarcinoma (OGA), pancreatic ductal adenocarcinoma (PDAC) and clinically challenging situations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oesophagogastric adenocarcinoma (OGA) (Experimental)
  Interventions: Diagnostic Test: [18F]AlF-FAPI-74 PET/CT
- Pancreatic ductal adenocarcinoma (PDAC) (Experimental)
  Interventions: Diagnostic Test: [18F]AlF-FAPI-74 PET/CT
- Clinically challenging situations (Experimental)
  Interventions: Diagnostic Test: [18F]AlF-FAPI-74 PET/CT

INTERVENTIONS:
Diagnostic Test: [18F]AlF-FAPI-74 PET/CT — A [18F]AlF-FAPI-74 PET/CT will be performed at the same site of the screening visit (UZ Leuven, UZ Gent or UZ Antwerpen). Subjects are required to be sober four hours before the scan. The patient will get an IV line, through which the [18F]AlF-FAPI-74 will be injected in one bolus (3,5 MBq/kg). After 60 minutes, the acquisition on the PET/CT scan will take place. The CT will be a low dose CT with oral contrast. After the scan, participants will be observed at the department in case of adverse events. During this time, the participant can fill in the PRO. The estimated duration of this visit is three hours. If the patient receives neo-adjuvant therapy, a second [18F]AlF-FAPI-74 PET/CT will be performed maximum one month before surgery. If the planned surgery gets postponed after the second [18F]AlF-FAPI-74 PET/CT has been performed, we will have the possibility to perform one additional (i.e. third) [18F]AlF-FAPI-74 PET/CT, before the final surgery.

SUMMARY:
The aim of the project is to demonstrate superior detection ratio of [18F]AlF-FAPI-74 PET/CT compared to [18F]FDG PET/CT or conventional imaging in treatment-naïve, newly diagnosed patients with oesophagogastric adenocarcinoma (clinical T1-4N0-3M0) and pancreatic ductal adenocarcinoma (clinical T1-4N0-2M0-1) and describe the clinical utility of [18F]AlF-FAPI-74 PET/CT in oncological patients with a clinically challenging situation.

ELIGIBILITY:
Inclusion Criteria OGA:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. Age 18 or older.
3. New histologic or cytologic proven diagnosis of oesophagogastric adenocarcinoma.
4. Patient underwent a [18F]FDG PET/CT.
5. TNM classification: cT1-4N0-3M0

Inclusion Criteria PDAC:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. Age 18 or older.
3. New histologic or cytologic proven diagnosis of pancreatic ductal adenocarcinoma.
4. Patient underwent a [18F]FDG PET/CT or conventional staging with CT or MRI.
5. TNM classification: cT1-4N0-2M0-1, with the exception of upfront resectable patients.

Inclusion Criteria Clinically challenging cohort:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. Age 18 or older.
3. Histologic or cytologic proven diagnosis of a malignancy.
4. Patient underwent a [18F]FDG PET/CT.
5. Unexplained symptoms, complaints, biochemical or imaging (scintigraphy, PET, CT, MR) findings.

Exclusion Criteria:

1. Participant is mentally or legally incapacitated, doesn't understand the study design or is not willing or capable to undergo all study-specific procedures.
2. Any disorder or condition, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial.
4. Female who is pregnant (urinary hCG test can be performed in case of doubt), breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive (with a relatively high Pearl Index: natural methods, minipill outside postpartum period, spermicides or condoms in monotherapy or no usage of contraception when sexually active are not accepted).
5. Participation in an interventional Trial with an investigational medicinal product (IMP) or device when the trial designs are not considered compatible by the study team.
6. Participation in a clinical scientific study in the last 12 months with a radiation exposure caused by the experimental procedures greater than 1 mSv.
7. Participant has a known hypersensitivity to [18F]AlF-FAPI-74 or the used excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective OGA: demonstrate superiority of [18F]AlF-FAPI-74 PET/CT over [18F]FDG PET/CT. | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Detection ratio for lymph node and distant metastases (combined).
Primary Objective PDAC: demonstrate superiority of [18F]AlF-FAPI-74 PET/CT over conventional imaging (CT or MRI) or [18F]FDG PET/CT (if available) | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Detection ratio for lymph node and distant metastases (combined).
Primary Objective Clinically Challenging Situation: demonstrate contribution of [18F]AlF-FAPI-74 PET/CT in this setting. | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Fraction of patients were scan was deemed contributory. This means:
  1. [18F]AlF-FAPI-74 identifies a lesion as malignant (true positive) with effective upstaging.
  2. [18F]AlF-FAPI-74 identifies a lesion as non-malignant (true negative) with effective downstaging.
  3. [18F]AlF-FAPI-74 can differentiate between a malignant or non-malignant lesion when there is doubt.
  4. Other implications that are deemed contributory by the treating physician.

SECONDARY OUTCOMES:
OGA & PDAC: Detection ratio for tumor detection | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  primary tumor alone; lymph nodes alone (N-staging); distant metastases alone (M-staging) and lymph node + distant metastases combined (with inclusion of patients without N- or M-lesions).
OGA & PDAC: specificity, positive and negative predictive value and accuracy | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Specificity, positive predictive value, negative predictive value, accuracy for lymph node and distant metastases (combined); for detection of primary tumor; for lymph nodes alone (N-staging); for distant metastases alone (M-staging).
OGA & PDAC: positive and negative likelihood ratios; diagnostic odds ratio. | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Positive and negative likelihood ratios; diagnostic odds ratio.
OGA & PDAC: semi-quantitative uptake measurements | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Semi-quantitative uptake measurements (maximal standardized uptake value (SUVmax), average SUV (SUVmean), peak SUV (SUVpeak) of tumoral lesions on [18F]AlF-FAPI-74 PET/CT and [18F]FDG PET/CT.
OGA & PDAC: tumor-to-background uptake values | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Tumor-to-background uptake values (TBR; SUV lesion divided by SUV background) for [18F]AlF-FAPI-74 PET/CT and [18F]FDG PET/CT, using following background organs: liver, lung, gluteus muscle, mediastinal bloodpool, bowel, bone marrow (L4 if no abnormal uptake).
OGA & PDAC: impact on TNM stage | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Impact on TNM stage of [18F]AlF-FAPI-74 PET/CT compared to full staging ([18F]FDG PET/CT and conventional imaging) and impact of [18F]AlF-FAPI-74 PET/CT compared to only conventional imaging-based staging.
OGA & PDAC: impact on clinical management | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Impact on clinical management.
OGA & PDAC: impact on potential radiation therapy plan | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Impact on potential radiation therapy plan.
OGA & PDAC: psychological impact | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Psychological impact on patient of [18F]AlF-FAPI-74 PET/CT procedure.
OGA & PDAC: reproducibility | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Intra- and interobserver reproducibility of both [18F]FDG and [18F]AlF-FAPI-74 PET/CT.
OGA & PDAC: adverse events | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Patient safety: adverse events of [18F]AlF-FAPI-74 PET/CT.
OGA & PDAC: evolution between baseline and end of neo-adjuvant treatment | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Evolution between baseline and end of neo-adjuvant treatment in patients with 2 [18F]AlF-FAPI-74 scans: (i) number of lesion; (ii) uptake; (iii) TBR; (iv) TNM score;(v) treatment plan based on scan.
OGA & PDAC: correlation with immunohistochemistry | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Correlation of [18F]AlF-FAPI-74 biodistribution with FAP tissue expression as measured by immunohistochemistry (IHC).
Subgroup analysis OGA: lymph node detection | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 1: Upfront resectable patients. Subgroup 2: Patients scheduled for neo-adjuvant therapy (mostly classified as locally advanced).
  Sensitivity, specificity, postivie predictive value, negative predictive value for lymph nodes.
Subgroup analysis OGA: impact on TNM stage | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 1: Upfront resectable patients. Subgroup 2: Patients scheduled for neo-adjuvant therapy (mostly classified as locally advanced).
  Impact on TNM stage of [18F]AlF-FAPI-74 PET/CT compared to [18F]FDG PET/CT-based stage.
Subgroup analysis OGA: evolution between baseline and end of neo-adjuvant treatment | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 2: Patients scheduled for neo-adjuvant therapy (mostly classified as locally advanced).
  Evolution between baseline and end of neo-adjuvant treatment in patients with 2 [18F]AlF-FAPI-74 scans: (i) number of lesion; (ii) uptake; (iii) TBR; (iv) TNM score; (v) treatment plan based on scan
Subgroup analysis OGA: correlation with pathology | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 2: Patients scheduled for neo-adjuvant therapy (mostly classified as locally advanced).
  Correlation of imaging parameters and their change with pathological assessment of resection specimen (pTNM stage, regression grade).
Subgroup analysis PDAC: tumor detection | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 1: Patients scheduled for neo-adjuvant therapy (mostly classified as borderline resectable or locally advanced).
  Subgroup 2: Metastatic patients. Sensitivity, specificity, positive predictive value, negative predictive value and accuracy for lymph nodes and distant metastases.
Subgroup analysis PDAC: impact on TNM stage | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 1: Patients scheduled for neo-adjuvant therapy (mostly classified as borderline resectable or locally advanced).
  Subgroup 2: Metastatic patients. Impact on TNM stage of [18F]AlF-FAPI-74 PET/CT compared to [18F]FDG PET/CT, CT or MRI-based stage.
Subgroup analysis PDAC: evolution between baseline and end of neo-adjuvant treatment | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 1: Patients scheduled for neo-adjuvant therapy (mostly classified as borderline resectable or locally advanced).
  Evolution between baseline and end of neo-adjuvant treatment in patients with 2 [18F]AlF-FAPI-74 scans: (i) number of lesion; (ii) uptake; (iii) TBR; (iv) TNM score; (v) treatment plan based on scan
Subgroup analysis PDAC: correlation with pathology | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 1: Patients scheduled for neo-adjuvant therapy (mostly classified as borderline resectable or locally advanced).
  Correlation of imaging parameters and their change with pathological assessment of resection specimen (pTNM stage, regression grade).
Subgroup analysis PDAC: association with survival | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Subgroup 2: Metastatic patients. Association between total tumor burden on [18F]AlF-FAPI-74 PET/CT and survival. Association between semi-quantitative uptake measurements (maximal standardized uptake value (SUVmax), average SUV (SUVmean), peak SUV (SUVpeak) of tumoral lesions on [18F]AlF-FAPI-74 PET/CT and survival.
Clinically Challenging Situation: detection rate | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Primary tumor/local recurrence, lymph node and distant metastases detection rate (compared to best value comparator) vs. [18F]FDG PET/CT.
Clinically Challenging Situation: semi-quantitative uptake measurements | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Semi-quantitative uptake measurements (maximal standardized uptake value (SUVmax), average SUV. (SUVmean), peak SUV (SUVpeak)) of tumoral lesions on [18F]AlF-FAPI-74 PET/CT and [18F]FDG PET/CT
Clinically Challenging Situation: tumor-to-background uptake values | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Tumor-to-background uptake values (SUV lesion divided by SUV background) on [18F]AlF-FAPI-74 PET/CT and [18F]FDG PET/CT, using following background organs: liver, lung, gluteus muscle, mediastinal bloodpool, bowel, bone marrow (L4 if no abnormal uptake).
Clinically Challenging Situation: impact on potential radiation therapy plan | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Impact on potential radiation therapy plan of [18F]AlF-FAPI-74 PET/CT vs. [18F]FDG PET/CT.
Clinically Challenging Situation: reproducibility | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Intra- and interobserver reproducibility.
Clinically Challenging Situation: adverse events | From enrollment to the end of the follow-up period (i.e. 12 months after first [18F]AlF-FAPI-74 PET/CT)
  Patient safety: adverse events.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - University Hospital Antwerp (UZA), Edegem
  - University Hospital Ghent, Ghent
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No